CLINICAL TRIAL: NCT02029547
Title: Evaluation of Computer-Based Training to Educate Japanese Physicians in the Methods of Interpreting Florbetapir (18F) PET Scans
Brief Title: Evaluation of Electronic Florbetapir (18F) Interpretation Training in Japanese Physicians
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-JPT01
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physician Readers (Experimental): Physician readers will interpret 60 Amyvid scans using qualitative analysis followed by the use of quantitation. No subjects will be exposed to florbetapir (18F) as part of this study.
  Interventions: Drug: Florbetapir (18F)

INTERVENTIONS:
Drug: Florbetapir (18F) — No Florbetapir (18F) will be administered in this study.
  Other Names: Florbetapir F 18; florbetapir; Amyvid; 18F-AV-45

SUMMARY:
This study is designed to validate the Japanese electronic florbetapir (18F) interpretation training program intended for post-approval implementation in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Japanese Society of Nuclear Medicine (JSNM) Positron Emission Tomography (PET) Certified Nuclear Medicine Physician
* Minimal hands-on experience and no formal training in the visual interpretation of florbetapir (18F) brain PET scans
* Minimal hands-on experience and no formal training in the quantitation of florbetapir (18F) brain PET scans

Exclusion Criteria:

* Prior hands-on experience or formal training in the visual interpretation and/or quantitation of florbetapir (18F) PET scans

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Inter Rater Reliability | Scan acquired 50-60 minutes post injection
  Measure of agreement among readers using a binary visual read method (amyloid positive/negative) calculated using Fleiss' kappa. All scans were read in a blinded fashion without access to clinical information.
Percent Agreement with Expert Panel | Scan acquired 50-60 minutes post-injection
  Individual reader scan results will be compared to the expert panel's consensus rating for each scan.

SECONDARY OUTCOMES:
Change in inter reader reliability after application of quantitation software | Scan acquired 50-60 minutes post injection
  Evaluate the percent change in inter reader reliability after implementation of quantitation analysis.
Change in agreement with expert panel | Scan acquired 50-60 minutes post-injection
  The percent change in individual reader agreement with the expert panel's consensus rating will determined after implementation of quantitation analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Tokyo, Japan